CLINICAL TRIAL: NCT00227955
Title: Maintenance Therapies in Recurrent Depression-Study I
Brief Title: Comparing Various Treatments for Achieving and Maintaining Remission of Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 871250
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Depression
Keywords: Major depression
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Imipramine; Interpersonal Psychotherapy

INTERVENTIONS:
Drug: Imipramine
Behavioral: Interpersonal Psychotherapy

SUMMARY:
This study will evaluate the effectiveness of five combinations of drug therapy and psychotherapy in maintaining remission of depression symptoms in people with recurrent major depression.

DETAILED DESCRIPTION:
Depression is a serious illness that can interfere with a person's ability to work, study, sleep, eat, and enjoy activities that once were pleasurable. It is characterized by several symptoms, such as the following: persistent sad, anxious, or "empty" mood; feelings of hopelessness or pessimism; and feelings of guilt, worthlessness, or helplessness. If left untreated, depression symptoms can last for years, and may worsen as time goes on. Even with treatment, however, it is possible for depression to recur. Remission is a main goal in the treatment of depression and it may be accomplished through various strategies. This study will evaluate the effectiveness of five combinations of treatments, including medication therapy and psychotherapy, in maintaining remission of depression symptoms.

All participants in this study will first be treated with imipramine for 7 to 11 months. Once remission of depression symptoms has been achieved and maintained for 20 weeks, participants will be randomly assigned to one of the following five maintenance treatments for 36 months: psychotherapy plus imipramine; psychotherapy plus placebo; psychotherapy alone; medication clinic treatment plus imipramine; or medication clinic treatment plus placebo. Assessments will be made at Weeks 12 and 20 and Months 7, 11, and 36, and will include the time it takes for depression symptoms to recur, as well as scores on depression and mania severity scales.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent major depression

Exclusion Criteria:

* Unstable medical illness
* Any other simultaneous psychiatric or medical illness of greater concern than depression (index episode of depression is not primary)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 1987-12; Study Completion 1993-12

PRIMARY OUTCOMES:
Time to recurrence of depression symptoms

SECONDARY OUTCOMES:
Measured at Months 7, 11, and 36: Score on the Raskin Depression and Mania Severity Scales

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Frank, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Cinic, Pittsburgh, Pennsylvania, United States